CLINICAL TRIAL: NCT04430348
Title: PTX35-001 A Phase I, First-in-Human, Dose-Escalation Study to Evaluate the Safety of the Monoclonal Antibody PTX-35 in Patients With Advanced Solid Tumors Refractory to Standard of Care
Brief Title: PTX-35 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Absence of immunological response
Sponsor: Pelican Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Heat Biologics (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PTX35-001
Record Dates: First submitted 2020-06-04; First posted 2020-06-12 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- PTX-35 Dose Level 1 (Experimental): Dose Level 1: PTX-35 0.01 mg/kg
  Interventions: Drug: PTX-35
- PTX-35 Dose Level 2 (Experimental): Dose Level 2: PTX-35 0.03 mg/kg
  Interventions: Drug: PTX-35
- PTX-35 Dose Level 3 (Experimental): Dose Level 3: PTX-35 0.10 mg/kg
  Interventions: Drug: PTX-35
- PTX-35 Dose Level 4 (Experimental): Dose Level 4: PTX-35 0.30 mg/kg
  Interventions: Drug: PTX-35
- PTX-35 Dose Level 5 (Experimental): Dose Level 5: PTX-35 1.0 mg/kg
  Interventions: Drug: PTX-35
- PTX-35 Dose Level 6 (Experimental): Dose Level 6: PTX-35 3.0 mg/kg
  Interventions: Drug: PTX-35

INTERVENTIONS:
Drug: PTX-35 — Monoclonal antibody PTX-35

SUMMARY:
A Phase I, First-in-Human, Dose-Escalation Study to Evaluate the Safety of the Monoclonal Antibody PTX-35 in Patients with Advanced Solid Tumors Refractory to Standard of Care

DETAILED DESCRIPTION:
This is an open-label, single arm, first-in-human, Phase I study of intravenous administration of PTX-35 to patients with advanced solid tumors refractory to, or ineligible for, or who refuse available SOC. Five escalating dose levels of PTX-35 will be explored using a traditional 3+3 design based on dose-limiting toxicities (DLTs) until optimal immunological dose (OID) or maximum tolerated dose (MTD) is established.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a patient must:

1. Be willing and have the capacity to sign the written informed consent form.
2. Be male or female of at least 18 years of age at the time of signing informed consent.
3. Have a documented diagnosis of metastatic or advanced, unresectable solid tumor disease. Patient must have progressed or recurred following standard of care (SOC) therapies, or are ineligible for, or who refuse other safe and effective SOC therapies, and whom the Investigator believes may benefit from experimental treatment with PTX-35.
4. Have an acceptable organ function, as defined below:

   1. Albumin ≥ 2.5 g/dL
   2. Total bilirubin < 3.0 × upper limit of normal (ULN), unless patient has Gilbert's syndrome
   3. Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3.0 × ULN, or

      * 5 × ULN in the case of liver metastases
   4. Calculated or measured creatinine clearance > 35 mL/minute per the Cockcroft-Gault formula
   5. Absolute neutrophil count ≥ 1,500/mm3
   6. Hemoglobin ≥ 9 g/dL
   7. Platelet count ≥ 100,000/mm3
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Have life expectancy of at least three months.
7. Patients, both females and males, of childbearing/reproductive potential must agree to use adequate contraception while included in the trial and for six months after the last treatment with PTX-35.

Exclusion Criteria:

In order to participate in this study, a patient must not:

1. Have received any systemic anticancer therapy including small molecules, chemotherapy, radiation therapy, monoclonal antibodies or any other experimental drug within 4 weeks of first dose of PTX-35. Adjuvant anti hormonal treatment(s) for prior breast cancer or prostate cancer are allowed. (Note: washout for palliative radiation therapy is 2 weeks).
2. Have clinically significant cardiac disease, including:

   1. Onset of unstable angina within 6 months of signing the Informed Consent Form (ICF).
   2. Acute myocardial infarction within 6 months of the signing the ICF.
   3. Known congestive heart failure (Grade III or IV as classified by the New York Heart Association); and/ or a known decreased cardiac ejection fraction (LVEF) of < 45%.
   4. Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥ 100 mmHg, despite optimal medical management.
3. Have known or clinically suspected leptomeningeal disease. Stable, previously treated metastases in the brain or spinal cord, are allowed as long as these are considered stable (by CT or MRI), and not requiring systemic corticosteroids.
4. Have a history of ≥ Grade 3 allergic reactions, or suspected allergy or intolerance to monoclonal antibody therapies.
5. Have a history of suspected cytokine release syndrome (CRS).
6. Have any known immunodeficiency disorders (testing not required).
7. Have received prior allogeneic stem cell transplant.
8. Have ongoing or current autoimmune disease. Permanent but stable and manageable immune related adverse events (irAE) from prior therapies are permissible, if prednisone equivalent corticosteroid use does not exceed 10 mg/day.
9. Have any other condition requiring concurrent systemic immunosuppressive therapy (other than allowable exceptions which do not exceed 10mg/day of prednisone/corticosteroid use).
10. Have clinically significant active viral, bacterial or fungal infection requiring:

    1. Intravenous treatment with antimicrobial therapy completed less than two weeks prior to first dose, or
    2. Oral treatment with antimicrobial therapy completed less than one week prior to first dose. Prophylactic treatment with antibiotics (e.g. for dental extractions) is allowed.
11. Have had major surgery (requiring general anesthesia or inpatient hospitalization) within four weeks before first administration of PTX-35.
12. Have had a known tetanus/diphtheria vaccine within the past 10 years.
13. Have known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least two years.
14. Have known previously untreated or symptomatic metastases in the brain or spinal cord requiring steroids. Patients with treated and stable CNS metastases may be enrolled after approval of the sponsor and/or Medical Monitor.
15. Have any other ongoing significant, uncontrolled medical condition in the opinion of the Investigator.
16. Have known positive serology for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C (except in cases of immunity after cured infection). Testing not required.
17. Have a history of substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the trial or evaluation of the trial result.
18. Be a female patient who is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W Tolcher, MD, Principal Investigator — Next Oncology
Locations (3):
- United States (3):
  - Providence Cancer Institute, Earle A. Chiles Research Institute, Portland, Oregon
  - NEXT Oncology Austin, Austin, Texas
  - Next Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTX-35 Dose Level 1 | PTX-35 Dose Level 2 | PTX-35 Dose Level 3 | PTX-35 Dose Level 4 | PTX-35 Dose Level 5 | PTX-35 Dose Level 6
Started | 3 | 3 | 4 | 3 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3 | 3 | 6
Not completed — Death | 3 | 2 | 2 | 2 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTX-35 Dose Level 1 | PTX-35 Dose Level 2 | PTX-35 Dose Level 3 | PTX-35 Dose Level 4 | PTX-35 Dose Level 5 | PTX-35 Dose Level 6 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6 | 22
Age, Continuous [Median (Full Range); unit: years] | 75 [67 to 76] | 68 [60 to 69] | 54 [39 to 73] | 76 [70 to 77] | 61 [47 to 79] | 60 [42 to 90] | 67.5 [39 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 2 | 3 | 3 | 14
  Male | 2 | 0 | 2 | 1 | 0 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 4 | 3 | 2 | 6 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 3 | 3 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Any Treatment-emergent Adverse Events (TEAEs) During the Trial
Description: TEAEs during the trial
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PTX-35 Dose Level 1 | PTX-35 Dose Level 2 | PTX-35 Dose Level 3 | PTX-35 Dose Level 4 | PTX-35 Dose Level 5 | PTX-35 Dose Level 6
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 6
Participants | 2 | 3 | 4 | 3 | 3 | 6

ADVERSE EVENTS:
Time Frame: At least 12 months
Arm/Group | PTX-35 Dose Level 1 | PTX-35 Dose Level 2 | PTX-35 Dose Level 3 | PTX-35 Dose Level 4 | PTX-35 Dose Level 5 | PTX-35 Dose Level 6
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 2/4 | 2/3 | 2/2 | 4/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4 | 2/3 | 2/3 | 2/6
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 4/4 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTX-35 Dose Level 1 (N=3) | PTX-35 Dose Level 2 (N=3) | PTX-35 Dose Level 3 (N=4) | PTX-35 Dose Level 4 (N=3) | PTX-35 Dose Level 5 (N=3) | PTX-35 Dose Level 6 (N=6)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestine obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTX-35 Dose Level 1 (N=3) | PTX-35 Dose Level 2 (N=3) | PTX-35 Dose Level 3 (N=4) | PTX-35 Dose Level 4 (N=3) | PTX-35 Dose Level 5 (N=3) | PTX-35 Dose Level 6 (N=6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement, Non-disclosure and Clinical Trial Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT04430348/Prot_SAP_000.pdf